CLINICAL TRIAL: NCT01752621
Title: Incidence and Late Prognosis of Acromegaly in Denmark From 1991 - 2010: Twenty Years of Medical Treatment
Brief Title: Epidemiology of Acromegaly in Denmark 1991-2010
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 3-3013-97/1/HKR; 11-88-37-29 (Other: data protection agency)
Record Dates: First submitted 2012-11-08; First posted 2012-12-19 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; mortality; morbidity; incidence; prevalence
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- acromegaly: patients with acromegaly
- comparison population: matched background population

SUMMARY:
Aim: To assess the incidence rate, morbidity and mortality of acromegaly in Denmark.

DETAILED DESCRIPTION:
Background: Acromegaly is a rare disease caused by GH hypersecretion from a pituitary adenoma. The annual incidence is estimated to be 3-5/million with a prevalence of 100 - 150/million. The incidence rate is however uncertain since no nationwide surveys exist. If left untreated or poorly controlled the condition is associated with progressive morbidity and an excess mortality. The primary treatment is surgery, which however only provides a cure rate of ≈ 50 -60% due to the size of the tumour. The second line treatment today is medical treatment with slow release formulations of somatostatin analogs (SA) and, more recently, a specific GH antagonist.

Accurate data on incidence rates and outcome of treatment are of obvious importance in order to provide optimal and evidence-based treatment for the disease. This is particularly relevant in light of the availability of new and effective treatment modalities such as the GH antagonist, the proper place of which in the treatment algorithm still remains controversial.

Denmark holds a unique position in terms of epidemiological studies due to the existence of well organized databases which include all its inhabitants. A recognised problem with epidemiological surveys from specialised centres is whether the figures are representative for the general population. A nationwide Danish study will profit from the fact that every Danish citizen holds a unique ID number that makes it easy to retrieve and combine pertinent data regarding health, disease and death from different registries. The investigators have previously used this for a landmark survey of another rare endocrine disease, i.e. Cushing's syndrome. This publication has been cited more than 100 times.

Aim: To assess the incidence rate, morbidity and mortality of acromegaly in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with acromegaly in years 1991-2010

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The entire danish population in the period 1991-2010 by means of national register
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Mortality of acromegaly | 3 years
  Mortality and morbidity of acromegaly (MRR)

SECONDARY OUTCOMES:
• Incidence of Acromegaly | 3 years
  • Incidence of Acromegaly
prevalence rates of Acromegaly | 3 years
  prevalence rates of Acromegaly

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto Jorgensen, professor, Study Director — MEA AUH
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Aarhus
  - Jakob Dal, Aarhus, Aarhus